CLINICAL TRIAL: NCT04931979
Title: Radiotherapy in Combination With Pembrolizumab in Patients With PSA Persistence or Biochemical Recurrence After Radical Prostatectomy Due to Prostate Cancer
Brief Title: SRT in Combination With Pembrolizumab in Patients With Recurrent Prostate Cancer After Radical Prostatectomy
Acronym: Pembro-SRT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. med. Christian Gratzke (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Christian Gratzke, Principal Investigator, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-3475-C51; 2021-001291-42 (EudraCT Number); P003141 (Other: Internal Protocol ID No.)
Record Dates: First submitted 2021-04-19; First posted 2021-06-18 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-11

CONDITIONS: Urologic Cancer; Biochemical Recurrence of Malignant Neoplasm of Prostate
Keywords: urologic cancer; biochemical recurrence of prostate-specific antigen; radical prostatectomy; pembrolizumab
MeSH Terms: conditions — Urologic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: The trial is designed as a phase II, open-label, monocentric, single-arm trial evaluating a combination therapy of pembrolizumab and salvage radiation therapy (SRT) in patients with biochemical recurrence (BCR) or persisting prostate-specific antigen (PSA) after radical prostatectomy (RP).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Pembrolizumab 200mg i.v. three-weekly in combination with salvage radiation therapy (SRT) according to standard of care
  Interventions: Drug: Pembrolizumab Injection [Keytruda]; Radiation: Salvage Radiation Therapy (SRT)

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Up to 17 cycles of pembrolizumab until disease progression, toxicity, death, or withdrawal of IC (whichever occurs first)
Radiation: Salvage Radiation Therapy (SRT) — SRT according to standard of care (SRT with at least 66 Gy)

SUMMARY:
To evaluate the efficacy and safety of a pembrolizumab therapy of pembrolizumab in combination with standard salvage radiation therapy (SRT) in patients with biochemical recurrence (BCR) of prostate-specific antigen (PSA) persistence after radical prostatectomy (RP).

DETAILED DESCRIPTION:
Current guidelines recommend a salvage radiation therapy (SRT) with at least 66 Gy as preferred treatment option in patients with biochemical recurrence (BCR) resp. PSA (prostate-specific antigen) persistence after radical prostatectomy (RP). The guideline recommendation is based on two non-randomized controlled trials that showed an improved cancer-specific survival and a better local tumor control. The optimal timing for a radiation therapy cannot be clearly defined by the available literature. A radiation therapy as early as possible with a PSA level <0,5 ng/ml seems to be beneficial. The guideline recommendation is based on two non-randomized controlled trials that showed an improved cancer-specific survival and a better local tumor control. A complete biochemical response is to be expected in approx. 60-70% of patients after 12 months.

The established imaging modality in patients with BCR used to be computed tomography of the abdomen and bone scintigraphy for the detection of skeletal lesions. The introduction of PSMA PET/CT (prostate-specific membrane antigen positron emission tomography combined with CT) has changed the imaging in patients with recurrent prostate cancer and several studies could show improved oncological results compared to patients undergoing standard treatment without positron emission tomography (PET) positive lesions with a 10% improvement in biochemical recurrence-free survival after 2 years.

Immunotherapy alone has not yet proven to be efficacious in prostate cancer as a monotherapy in smaller studies. Several trials could show that the combination of the immunotherapy and radiation therapy has the potential to provide a synergistic effect in treating genitourinary malignancies, whereas more studies are needed to uncover the exact underlying mechanism. In brief, radiation therapy of the location of recurrence increases the tumor´s immunogenic potential and a systemic immunological reaction is initiated that leads to an increased activity of the immune system against tumor tissue (abscopal effect). Lately several trials have been evaluating a possible synergistic effect with tolerable side-effects. A trial combining those two treatment regimens in the early treatment of prostate cancer recurrence is not available up to date.

The clinical benefit of concomitant androgen deprivation therapy (ADT) is controversial and literature failed to show a clear overall survival benefit for all patients. Several retrospective trials have been evaluating a concomitant ADT and for patients with risk factors like suspicious lymph-nodes in staging diagnostics. Several studies have been evaluating the effect of concomitant ADT though. Shipley et al. could show the addition of 24 months of bicalutamide to SRT resulted in significantly higher rates of long-term overall survival. However, sub-group analyses revealed that this effect counts mainly for patients with PSA of >0.7 ng/ml before SRT. The GETUG-AFU trial did not find any survival benefit for short term (6 months) ADT additionally to SRT. However, a significant benefit in progression-free survival after 120 months of follow-up time was reported. A combination therapy of pembrolizumab and radiation therapy has not been evaluated before in this patient population. The investigators hypothesize that this combination is more effective than radiation therapy alone due to a radiogenic triggered immunomodulation which increases the anti-tumor effect of pembrolizumab. For patients with BCR or PSA persistence after RP no such treatment regimen has been tested yet.

ELIGIBILITY:
Inclusion criteria:

1. Male patients who are at least 18 years of age on the day of signing informed consent
2. Histologically confirmed diagnosis of an adenocarcinoma of the prostate and a BCR or PSA persistence after RP
3. Histology of the RP specimen needs to fulfill the following criteria: adenocarcinoma of the prostate, Gleason score 7-10; pNX or pN0 or pN1 (max. 2 lymph nodes involved)
4. Imaging within 50 days prior to study inclusion is mandatory (patient registration) ([68Ga] or [18F] PSMA PET-CT as standard imaging modality, alternatively CT abdomen and full-body bone scan)
5. PSA value between ≥0.2 and ≤1.0 ng/ml measured at least six weeks postoperatively
6. The patients agree not to undergo testicular sperm extraction for at least 90 days after the last administration of pembrolizumab. (Due to prior surgical removal of the prostate no contraception is necessary.)
7. Written informed consent obtained according to international guidelines and local law
8. Patients further having an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
9. Patients with adequate organ function as defined in clinical trial protocol (CTP) (Section 4)

Exclusion criteria:

1. Prior-therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
2. Prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to registration (like neo-adjuvant androgen deprivation therapy (ADT), secondary hormone ablation or taxan-based chemotherapy).
3. Prior radiotherapy within 4 weeks before start of study medication. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
4. Distant metastases or suspicious lymph nodes outside the lower pelvis in imaging with PSMA PET-CT are to be excluded (patients with PET positive bone lesions that are morphologically not clearly suspicious of metastases and would not change clinical practice can be included).
5. Adverse histology of RP specimen (e.g. neuroendocrine or small cell)
6. Any vaccination with live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study medication. Administration of killed vaccines is allowed.
7. Currently or previously participating in a study of an investigational product within 4 weeks prior to the first dose of study medication.
8. Diagnosis of immunodeficiency, chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication.
9. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
10. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
11. Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
12. Active autoimmune disease that required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
13. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or currently pneumonitis/ interstitial lung disease
14. Active infection requiring systemic therapy.
15. History of Human Immunodeficiency Virus (HIV) infection.
16. History of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as Hepatitis C virus (HCV) RNA is detected) infection. No testing is required.
17. History of active TB (Bacillus Tuberculosis).
18. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the investigator.
19. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
20. History of allogeneic tissue/solid organ transplantation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Complete biochemical response | at week 60 (+/- weeks) after start of treatment
  number of patients with complete biochemical response defined as a PSA level below limit of detection.
  Patients will be counted as a responder with respect to the primary endpoint, if the PSA level is below the limit of detection at week 60 (± 2 weeks) after start of trial treatment. Patients will be counted as a non-responder with respect to the primary endpoint, if the PSA level is above the limit of detection at week 60 (± 2 weeks).

SECONDARY OUTCOMES:
Radiographic progression-free survival | at week 60 (+/- 2 weeks) after start of treatment
  The probability of radiographic progession-free survival at week 60 (+/- 2 weeks) after start of treatment will be estimated as the number of patients who are alive and progression-free divided by the total number of treated patients.

OTHER OUTCOMES:
PSA-nadir level | lowest PSA level during pembrolizumab administration (49 weeks)
  The PSA-nadir is defined as the lowest PSA-level measured after start of pembrolizumab administration.
Time to PSA-nadir (TNN) | from start of trial treatment (visit 1/cycle 1) to lowest PSA level (up to 17 visits/ cycles of trial treatment during 49 weeks)
  The time to PSA-nadir is defined as the time from start of pembrolizumab administration to this time point.
Duration of pembrolizumab exposure | from start of pembrolizumab administration (cycle 1/visit 1) to up to visit /cycle 17 during 49 weeks for each patient, each cycle is 21 days
  Number of administered pembrolizumab cycles.
Dose of pembrolizumab | from start of pembrolizumab administration (cycle 1/visit 1) to up to visit /cycle 17 during 49 weeks for each patient, each cycle is 21 days
  Cumulative dose as sum of all pembrolizumab doses given.
Dose intensity of pembrolizumab | from start of pembrolizumab administration (cycle 1/visit 1) to up to visit /cycle 17 during 49 weeks for each patient, each cycle is 21 days
  Cumulative dose as sum of all pembrolizumab doses given divided by the time under pembrolizumab treatment (last date minus first date of administration).
Dose changes of pembrolizumab | from start of pembrolizumab administration (cycle 1/visit 1) to up to visit /cycle 17 during 49 weeks for each patient, each cycle is 21 days
  Number of patients with dose change of pembrolizumab along with reasons for dose change.
Dose interruptions of pembrolizumab | from start of pembrolizumab administration (cycle 1/visit 1) to up to visit /cycle 17 during 49 weeks for each patient, each cycle is 21 days
  Number of patients with interruptions of pembrolizumab administration along with reasons for dose interruptions.
Dosage of subsequent Androgen Deprivation Therapy (ADT) in high-risk patients (cN+ in imaging or PSA >0.7 ng/ml at screening) | Month 6 after start of pembroblizumab administration to end of study (week 72)
  Cumulative dose of ADT after month 6 after start of pembrolizumab administration.
Time to initiation of subsequent Androgen Deprivation Therapy (ADT) in high-risk patients (cN+ in imaging or PSA >0.7 ng/ml at screening) | Month 6 after start of pembroblizumab administration to end of study (week 72)
  Time from month 6 after start of pembrolizumab administration to start of ADT.
Dosage of Androgen Deprivation Therapy (ADT) in low-risk patients | Start of pembroblizumab administration to end of study
  Cumulative dose of ADT after start of pembrolizumab administration.
Time to initiation of Androgen Deprivation Therapy (ADT) in low-risk patients | Start of pembroblizumab administration to end of study (week 72)
  Time from start of pembrolizumab administration to start of ADT.
Functional assessment of cancer therapy - prostate cancer (FACT-P questionnaire, 4.0) | week 1, week 16, week 49, week 60
  Quality of life of patients will be evaluated using the Functional assessment of cancer therapy - prostate cancer (FACT-P questionnaire. The scoring and the analysis of the total score and the subscale scores will be performed according to the scoring manual available from www.facit.org.
  Minimum value: 0, Maximum value (FACT-P Trial Outcome Index, TOI): 104, Maximum value (FACT-G total score): 108, Maximum value (FACT-P total score): 156, High score indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gratzke, Prof. Dr., Principal Investigator — University Medical Center - University of Freiburg, Clinical of Urology
Locations (1):
- Clinic of Urology, Medical Center - University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No